CLINICAL TRIAL: NCT05635240
Title: Chronic Anterior Shoulder Instability in the Military
Acronym: EPAULUX
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PPRC13; 2022-A02091-42 (Other: IDRCB)
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview / questionnaires — At each of the 4 visits, the participant will have to answer several questions regarding trauma-related data, employment and sport practice.

SUMMARY:
Anterior shoulder instability is a chronic condition that occurs after an anteromedial dislocation. Its prevalence is high in athletes but has been little studied in the armed forces. In general, patients with a first episode of dislocation have a 1 in 2 chance of experiencing at least one recurrence. The more recurrences there are, the more damage there is to the joint and the greater the disability for the patient. The decree determining the medical aptitude of military personnel emphasizes the need to have recourse to a specialized consultation to determine the classification of the soldier after a first episode of dislocation. In the absence of data collected specifically in the military population, classification is based on the surgeon's experience and extrapolation of results obtained in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Military member with a first episode of true anterior glenohumeral shoulder dislocation,
* Male or female,
* Major,
* Having a sufficient level of reading/writing of the French language,
* Did not object to participating in the study.

Exclusion Criteria:

* Patient with a history of homolateral shoulder dislocation or surgery on the affected shoulder,
* Collagen disease confirmed by genetic testing,
* Inflammatory arthropathy,
* History of rotator cuff injury,
* Insufficient French reading/writing skills,
* Under legal protection,
* Objection to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of French military member with a first episode of true anterior glenohumeral shoulder dislocation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a new episode of true anterior glenohumeral shoulder dislocation or subluxation 1 year after the initial dislocation. | Through study completion (72 months)
  A true anterior glenohumeral shoulder dislocation is defined as a dislocation requiring reduction.
  Dislocation and subluxation will have to be objectified by medical examination

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Direction Médicale des Forces, Tours

IPD SHARING:
Plan to Share IPD: Undecided